CLINICAL TRIAL: NCT07295444
Title: A Clinical Study Evaluating the Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for Participants With Mild Depressive Disorder Comorbid With Anxiety Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRD-NX-KN-001
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Mild Depressive Disorder Comorbid With Anxiety Disorder
Keywords: Depressive Anxiety herbal capsules efficiency

STUDY DESIGN:
Masking Description: pharmacy administrator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Clinical Study Evaluating the Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for P (Experimental): Mild Depressive Disorder Comorbid With Anxiety Disorder
  Interventions: Dietary Supplement: A Clinical Study Evaluating the Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for Participants With Mild Depressive Disorder Comorbid With Anxiety Disorder

INTERVENTIONS:
Dietary Supplement: A Clinical Study Evaluating the Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for Participants With Mild Depressive Disorder Comorbid With Anxiety Disorder — A Clinical Study Evaluating the Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for Participants With Mild Depressive Disorder Comorbid With Anxiety Disorder

SUMMARY:
The incidence of Mild Depressive Disorder Comorbid With Anxiety Disorder is dramatically increasing. dietary supplements may show better efficiency and less side effect.Here investigators intend to assess Efficacy and Safety of CreNeuriS CNS Herbal Nutrition Capsules for Participants With Mild Depressive Disorder Comorbid With Anxiety Disorder.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, open-label, self-controlled clinical trial evaluating the efficacy and safety of CreNeuroS CNS Herbal Nutrition Capsules (CreNeuroS CNS Herbal Calm Capsules) in improving mild depressive disorder comorbid with anxiety disorder. The study plans to enroll a total of 30 participants, aged 18-65 years. Eligible participants will be screened and enrolled, stratified by age at 45 years. All participants will take the Herbal Calm Capsules twice daily, morning and evening, two capsules each time, continuously for 42 days, during which efficacy and safety will be assessed.

ELIGIBILITY:
Inclusion Criteria: 1. Age between 18 and 65 years old (including 18 and 65); 2. Diagnosed with depression according to the Mini International Neuropsychiatric Interview (MINI) and the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); Hamilton Depression Rating Scale (HAMD-17) score between 8 and 17 (inclusive); 3. Diagnosed with anxiety according to the Mini International Neuropsychiatric Interview (MINI) and the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); Hamilton Anxiety Rating Scale (HAMA) score between 14 and 20 (inclusive); 4. Possess basic comprehension and communication skills and be able to complete assessments independently or under guidance; 5. Fully understand and sign the informed consent form; 6. The subject commits to having no plans for conception or sperm/egg donation from the time of signing the informed consent until 3 months after the last dose of medication, and voluntarily agrees to strictly use one or more contraceptive measures (such as intrauterine device, condom).

Exclusion Criteria:

1. History of epilepsy, schizophrenia, bipolar and related disorders, intellectual disability, cognitive impairment, or any other neurological or psychiatric disorder that the investigator believes could affect the subject's safety or interfere with study assessments; 2. History of severe cardiovascular diseases meeting any of the following criteria:

1. Heart failure (New York Heart Association functional class ≥ III);
2. Unstable angina within the past 6 months;
3. Any arrhythmia requiring treatment;
4. QTc interval prolongation considered clinically significant by the investigator (reference range: men > 450 ms, women > 470 ms) (Note: QTc interval must be calculated according to Fridericia's formula);
5. Acute myocardial infarction or interventional procedure within the past month. 3. History of severe gastrointestinal diseases, such as active ulcers or gastrointestinal bleeding; 4. History of severe respiratory diseases, such as chronic obstructive pulmonary disease, cor pulmonale, pulmonary interstitial fibrosis, etc.; 5. Hypertension that is not well controlled by medication: systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg during the screening period. If the first measurement exceeds the limit, it can be repeated after at least 5 minutes on the same day. If three measurements still do not meet the criteria, the subject is ineligible; 6. Clinically diagnosed cerebrovascular accident or intracranial hemorrhage within 6 months; 7. History of moderate to severe sleep apnea, circadian rhythm sleep disorders, narcolepsy, restless legs syndrome, or sleep disorders secondary to other diseases; 8. History of complex sleep behaviors, such as previous episodes of driving, eating, or making phone calls during sleep; 9. Anxiety and/or depressive disorders, or insomnia requiring drug or other interventions during the trial; 10. Exclusion during screening if any of the following abnormalities are present:

1) Platelets (PLT) < 100 × 10^9/L, or hemoglobin (Hgb) < 90 g/L; 2) Liver function: AST or ALT > 3 × ULN, TBIL > 2 × ULN; 3) Renal function: serum creatinine > 2 × ULN. 11. History of severe allergic reactions (e.g., anaphylactic shock, laryngeal edema, severe bronchospasm); 12. High risk of suicide: suicide attempt within 1 year prior to screening; suicidal or self-harm behavior during screening; HAMD-17 item 3 (suicide) score ≥ 3; 13. History of abuse or addiction to relevant psychiatric medications; 14. Pregnant or breastfeeding women; 15. Participation in another drug clinical trial within 1 month prior to screening; 16. Any disease or condition that the investigator believes makes the subject unsuitable for participation in the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
HAMD-17 assessment chart | six weeks
  HAMD-17 assessment comparison between baseline and six weeks later
HAMD-17 assessment comparison between baseline and six weeks later | 6 weeks
  HAMD-17 assessment comparison between baseline and six weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- Second affiliated hospital of nanchang university, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No